CLINICAL TRIAL: NCT04529590
Title: Precise Treatment of Prediabetes and Stage 1 Hypertension
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-212
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
Keywords: 130-139/80-89 mmHg; all-cause mortality; cardiovascular mortality; glucose metabolism; Chinese
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10 ml serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with cardiovascular events after 18 years: Analyzing metabolic markers screened and optimized by multivariate statistical with plasma metabolic profiles from peripheral blood samples of different groups.
  Positive patients' samples will be collected at baseline.
- Patients without cardiovascular events after 18 years: For negative patients' samples will be collected at baseline as negative control.

SUMMARY:
To identify the occurrence of diabetes, hypertension, cardiovascular and cerebrovascular events and all-cause death in patients with baseline prediabetes and stage1 hypertension after 18 years follow up. To identify whether one or several metabolites can be used as serum markers to judge the prognosis of patients with prediabetes and stage1 hypertension, and to establish the evaluation model of metabolites for the prognosis.

DETAILED DESCRIPTION:
To identify the occurrence of diabetes, hypertension, cardiovascular and cerebrovascular events and all-cause death in patients with baseline prediabetes and stage1 hypertension after18 years follow up, then explore the role of risk factors. After assessing the association between BP categories and all-cause mortality and cardiovascular mortality, to analyze the risk for all-cause and cardiovascular mortality by blood glucose categories and BP categories combined by using multiple Cox regression analysis. To analyze the corresponding incidence of all-cause mortality per 1,000 person-years for the BP<130/80 mmHg, 130-139/80-89 mmHg, and ≥140/90 mmHg or treated groups respectively after adjusting for age, sex, and other factors. To identify the associations between cardiovascular mortality and BP categories alone or combined with blood glucose categories were consistent with that of all-cause mortality.

To identify relative metabolic molecular biomarker panel detected by mass spectrometry in blood samples correlating with efficacy in prediabetes and stage 1 hypertension among Chinese adults. Compare the plasma metabolic profiles of different groups and the metabolic markers were screened and optimized by multivariate statistical analysis, logistic regression analysis and receiver operating characteristic (ROC) curve analysis.

To determine whether one or several metabolites can be used as serum markers to judge the prognosis of patients with prediabetes and stage1 hypertension, and to establish the evaluation model of metabolites for the prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. aged from 18-76 years old
2. lived in Shanghai Pingliang community for 20 years
3. all participants' blood pressures are at baseline

Exclusion Criteria:

1. aged <18 years old or > 76 years old
2. with second primary malignant diseases. 3. other situations assessed by investigator can disturb quality control of the investigation.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female participants ages 18-76 years from the Pingliang community was conducted from November 2002 to January 2003. At baseline, all participants underwent physical examination and were interviewed with standardized questionnaires.
Sampling Method: Probability Sample
Enrollment: 2004 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of nonfatal myocardial infarction | 24 months
  The diagnosis of myocardial infarction includes clinical manifestations (symptoms and signs), measurement of cardiac biomarkers and ECG interpretation; myocardial infarction occurred during surgery / operation and myocardial infarction terminated due to thrombolytic therapy. According to the available data, the outcome evaluator will classify myocardial infarction into three categories: definite, probable and possible. All three types of myocardial infarction were included in the main outcome. Stroke can be judged based on all available data, including symptoms and signs, brain and large vessel imaging, and cardiac examinations such as echocardiography.
Rate of nonfatal stroke | 24 months
  Stroke can be divided into ischemic stroke, subarachnoid hemorrhage, cerebral parenchymal hemorrhage, other hemorrhage, other types or unknown types.
Rate of heart failure | 24 months
  Heart failure is defined as a clinical syndrome characterized by a variety of symptoms and signs of cardiac decompensation / cardiac pump insufficiency that are hospitalized or require infusion in the emergency room.
Rate of cardiovascular death | 24 months
  Cardiovascular death includes stroke, coronary heart disease, heart failure or other forms of cardiovascular disease (such as abdominal aortic aneurysm rupture, arrhythmia, etc.).

SECONDARY OUTCOMES:
Rate of major cardiovascular event composite endpoint | 24 months
  Macrovascular complication outcome: Stroke; Coronary heart disease:, coronary heart disease causes of death;Emergency treatment or hospitalization of heart failure; Cardiovascular death; All-cause death; Cognitive decline; Health-related quality of life.
  Macrovascular complication outcome: Stroke; Coronary heart disease:, coronary heart disease causes of death;Emergency treatment or hospitalization of heart failure; Cardiovascular death; All-cause death; Cognitive decline; Health-related quality of life.
Rate of all-cause death | 24 months
  all-cause death

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China